CLINICAL TRIAL: NCT05930782
Title: A Randomized, Open Label, Two-part, Parallel-group, Phase I Study to Evaluate the Pharmacokinetics of Piperaquine Oral Dispersible Granules Formulation Compared to Piperaquine Hard Tablets Administered as a Single Dose in Fasting Condition (Part 1) and of Piperaquine Oral Dispersible Granules Formulation Administered as Single Dose in Various Fed States (Part 2) in Healthy Adult Participants
Brief Title: Piperaquine Granule Formulation Relative Bioavailability and Food Effect Study in Healthy Volunteers.
Acronym: PedPQP(BA/FE)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MMV_SMC_22_01
Record Dates: First submitted 2023-06-26; First posted 2023-07-05 (Actual); Results first posted 2025-03-06 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Malaria
Keywords: Pharmacokinetics; Malaria prevention; Bioavailability; Malaria; Food effect; Oral granule formulation
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Intervention Model Description: Part 1: PQP tablet / dispersible granule administered in fasting condition of at least 10 hours.
  * Group 1: PQP hard tablet, 320 mg (N=12)
  * Group 2: PQP dispersible granule, 320 mg (N=12)
  Transition to Part 2:
  To minimize the risk to healthy participants, a decision on transitioning from Part 1 to Part 2, will be taken by the Safety Review Committee (SRC), based on the safety and preliminary PK interim report of the granule formulation, compared to the PQP hard tablet, with safety data obtained up to Day 15 and PK data obtained up to Day 8. If necessary, doses may be readjusted for the Part 2 to assess the food effect.
  Part 2: PQP dispersible granule administered in fed conditions (planned as 320 mg)
  * Group 3: High-fat meal (N=12)
  * Group 4: Low-fat meal representative of African diet (N=12)
  * Group 5: Whole milk 250 ml (N=12)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Part 1 (Fasted): Group 1: Piperaquine hard tablets (Active Comparator): Participants received a single oral dose of Piperaquine hard tablets 320mg (administered in fasting condition of at least 10 hours) (N=12)
  Piperaquine: Piperaquine tetraphosphate hard tablets 320mg
  Interventions: Drug: Piperaquine Tetraphosphate uncoated tablets
- Part 1 (Fasted): Group 2: Piperaquine dispersible granules (Experimental): Participants received a single oral dose of Piperaquine dispersible granule 320mg (administered in fasting condition of at least 10 hours) (N=12)
  Piperaquine: Piperaquine tetraphosphate dispersible granules 320mg
  Interventions: Drug: Piperaquine Tetraphosphate dispersible granules
- Part 2 (Fed): Group 3: Piperaquine dispersible granules (Experimental): Participants received a single oral dose of Piperaquine dispersible granule 320mg administered with a high-fat meal (N=12)
  Piperaquine: Piperaquine tetraphosphate dispersible granules 320mg
  Interventions: Drug: Piperaquine Tetraphosphate dispersible granules
- Part 2 (Fed): Group 4: Piperaquine dispersible granules (Experimental): Participants received a single oral dose of Piperaquine dispersible granule 320mg administered with a low-fat meal representative of African diet. (N=12)
  Piperaquine: Piperaquine tetraphosphate dispersible granules 320mg
  Interventions: Drug: Piperaquine Tetraphosphate dispersible granules
- Part 2 (Fed): Group 5: Piperaquine dispersible granules (Experimental): Participants received a single oral dose of Piperaquine dispersible granule 320mg administered with whole milk (250ml) (N=12)
  Piperaquine: Piperaquine tetraphosphate dispersible granules 320mg
  Interventions: Drug: Piperaquine Tetraphosphate dispersible granules

INTERVENTIONS:
Drug: Piperaquine Tetraphosphate uncoated tablets — Piperaquine tetraphosphate hard tablet 320 mg; single dose (320 mg) given orally with 240 ml of water
  Arms: Part 1 (Fasted): Group 1: Piperaquine hard tablets
Drug: Piperaquine Tetraphosphate dispersible granules — Piperaquine tetraphosphate dispersible granules 320 mg dose equivalent dispersed in 25 ml of water; single dose (320 mg) given orally
  Arms: Part 1 (Fasted): Group 2: Piperaquine dispersible granules; Part 2 (Fed): Group 3: Piperaquine dispersible granules; Part 2 (Fed): Group 4: Piperaquine dispersible granules; Part 2 (Fed): Group 5: Piperaquine dispersible granules

SUMMARY:
This trial aims to characterise the pharmacokinetic (PK) profile and estimate drug exposure of a single oral dose of piperaquine (PQP) in a dispersible granule formulation compared to the PQP hard tablet formulation in the fasted state (Part 1), to advise the selection of dose when the PQP granule formulation is administered in a fed state in healthy adult participants. Part 2 will assess the effect on different types of meal composition on the PK of a single dose of PQP granule formulation in healthy adult participants.

DETAILED DESCRIPTION:
Adult participants who give written informed consent will be screened within 45 days to determine their eligibility before entering the trial on Day -1. The trial will initially establish the pharmacokinetic (PK) profile and estimated drug exposure of a single oral dose of PQP in a dispersible granule formulation compared to the PQP hard tablet formulation in the fasted state (Part 1). In the second study part, and based on the PK results of Part 1, it is intended to administer the same dose level of 320 mg PQP dispersible granules concomitant with different fed conditions. However, if from Part 1 of the study it is shown that PQP dispersible granules formulation provides a significant improvement in Cmax values in the fasted state, this dose level may be adjusted for Part 2, in order to take into account a potential 3-fold increase in exposure which is the observed food effect when film-coated tablets (Eurartesim®) are administered with a high fat/high calorie meal. Such dose adjustment will be based on the safety and preliminary PK interim results of the granule formulation in the fasted state. The PQP dose selected in Part 2 (as dispersible granules formulation) will take into account a 3-fold factor increase in exposure when administered with food (see above) with such predicted exposure in the presence of food being not higher than after the administration of 960 mg PQP in tablet of Eurartesim® in adult subjects dosed in fasting conditions. Furthermore, sufficient data will be available to address key questions on both, safety and PK parameters to enable the review and recommendation by the SRC for the optimal dose of the granule formulation to be administered in Part 2.

ELIGIBILITY:
Inclusion Criteria:

Participants must fulfil all of the following criteria to be eligible for enrolment in this trial:

1. Female or Male aged ≥18 years to ≤55 years at the date of signing informed consent.
2. Ability to provide written, personally signed, and dated informed consent to participate in the trial, in accordance with the ICH Good Clinical Practice (GCP) and applicable regulations, before any trial-related procedures.
3. An understanding, ability, and willingness to fully comply with trial procedures and restrictions.
4. Female participants must agree to follow contraceptive requirements as indicated in Section 13.2.2, from at least 30 days prior to first dosage to 16 weeks after last dosage.
5. Agrees not to donate sperm or ova from the time of the first administration of trial medication until twelve weeks after the end of the systemic exposure of the trial drug.
6. Participants must have a body weight of 50 kg or greater and a BMI between 18.0 kg/m² - 30.0 kg/m² (inclusive) at screening.
7. Satisfactory medical assessment with no clinically significant or relevant abnormalities as determined by; medical history, physical examination, vital signs, 12-lead electrocardiogram (ECG) and clinical laboratory evaluation that is reasonably likely to interfere with the participant's participation in or ability to complete the trial as assessed by the Investigator.

Exclusion Criteria:

Participants will be excluded from enrolment in this trial if they fulfil any of the criteria below:

1. Prior screen failure or randomisation in this trial. NOTE: Participants who initially failed due to temporary non-medically significant issues are eligible for re-screening once the cause has resolved.
2. Female participant who is pregnant (from history, examination or confirmed by a positive serum pregnancy test at screening and/or on Day -1) or breastfeeding.
3. Male participants with a female partner(s) who is (are) pregnant or lactating at screening and/or on Day -1, or is (are) expected to be during the trial period.
4. Has a mental incapacity or language barriers precluding adequate understanding, co-operation, or compliance with the trial requirements.
5. Unable or unwilling to follow a standardised diet and meal schedule or unable to fast, as required during the trial.
6. Has milk intolerance.
7. Unable to swallow tablets.
8. Has veins on either arm that are unsuitable for intravenous puncture or cannulation (e.g., veins that are difficult to locate, or a tendency to rupture during puncture).
9. Known or suspected intolerance or hypersensitivity to the investigational products, any closely related compound, or any of the stated ingredients.
10. History of significant allergic reaction (e.g., anaphylaxis, angioedema) to any product (food, pharmaceutical, etc) but excluding untreated, asymptomatic, seasonal allergies.
11. Donated blood or blood products (excluding plasma) within 90 days prior to trial medication administration.
12. Has received or plans to receive a COVID-19 vaccination within two weeks before to one week after trial last visit.
13. Treated with medication containing PQP within 90 days or five half-lives preceding the dose of trial medication (whichever is the longer).
14. Ingested herbal remedies or dietary supplements containing St. John's Wort in the 30 days before the planned Day 1 of the dosing Part.
15. Taking medicinal products that are known to prolong the QTc interval (see http://www.crediblemeds.org/). An up-to-date list will be in the study specific manual.
16. Use of any medication that is either a moderate or strong inhibitor or inducer of CYP3A4 within 30 days or five half-lives (whichever is longer) prior to the planned day of dosing (see Drug Development and Drug Interactions, Table of Substrates, Inhibitors and Inducers, FDA). Anup to date list will be in the study specific manual.
17. Use of any other prescription medication (excluding hormonal contraception and hormone replacement therapy) within 14 days or ten half-lives (whichever is longer) prior to Day 1 of the dosing Part that the Investigator judges is likely to interfere with the trial or pose an additional risk in participating.
18. Use of any over-the-counter medication (including multivitamin, herbal, or homeopathic preparations; excluding paracetamol - up to 3 g of paracetamol per day permitted while participants are in-house, whereas while participants are outpatients a maximum of 1 g paracetamol per day will be allowed) during the seven days or ten half-lives of the drug (whichever is longer) prior to Day 1 of the dosing Part, that the Investigator judges is likely to interfere with the trial or pose an additional risk in participating.
19. Ingested any poppy seeds within the 24 hours prior to screening or admission.
20. Current use of tobacco in any form (e.g., smoking or chewing) or other nicotine-containing products in any form (e.g., gum, patch, electronic cigarettes).
21. History or clinical evidence of substance and/or alcohol abuse within the two years before screening. Alcohol abuse is defined as regular weekly intake of more than 14 units (for both males and females).
22. Participants must have not consumed other substances known to be potent inhibitors or inducers of CYP34A system such as grapefruit or cranberry juice containing products in the 30 days before the planned IMP administration.
23. Any history of seizures, epilepsy, photosensitivity or documented retinopathy.
24. The history or presence of any of the following cardiac conditions: known structural cardiac abnormalities; family history of long QT syndrome; cardiac syncope or recurrent, idiopathic syncope; exercise related clinically significant cardiac events.
25. Has vital signs consistently outside of the normal range at screening or Day-1.
26. Any clinically significant abnormalities in rhythm, conduction or morphology of resting ECG or clinically important abnormalities that may interfere with the interpretation of QTc interval changes. This includes participants with any of the following (at screening or Day -1):

    * sinus node dysfunction
    * clinically significant PR (PQ) interval prolongation (>220ms)
    * second- or third-degree atrioventricular (AV) block
    * sustained cardiac arrhythmia's including (but not limited to) atrial fibrillation or supraventricular tachycardia, or any symptomatic arrhythmia, with the exception of isolated extra-systoles
    * abnormal T-wave morphology which may impact on the QT/QTc assessment
    * QT interval corrected using the Fridericia's formula (QTcF) >450 ms
    * any other ECG abnormalities in the standard 12-lead ECG or an equivalent assessment which in the opinion of the Investigator will interfere with the ECG analysis
    * Participants with borderline abnormalities may be included if the deviations do not pose a safety risk, and if agreed between the appointed cardiologist and the PI.
27. Positive test results for alcohol or drugs of abuse at screening or Day -1.
28. Electrolyte imbalances, particularly results that are out of reference intervals for potassium, calcium or magnesium.
29. Has a positive test for Hepatitis B surface Antigen (HBsAg), Hepatitis C Antibody (HCV Ab), or Human Immunodeficiency Virus Antibody (HIV Ab) at screening.
30. Presence of malaria parasites by blood smear.
31. Has total bilirubin, ALT or AST consistently >upper limit of normal (ULN) at screening (up to two repeats may be taken during the screening period; participants may be included if two out of the three total results are ≤ULN), or has total bilirubin >ULN on Day -1 (mild variations from baseline may be allowed if considered not clinically significant by the Investigator).
32. Has a haemoglobin, platelet count, total white blood cell count, lymphocyte or monocyte count < lower limit of normal (LLN) (up to two repeats may be taken during the screening period and on Day -1 (participants may be included if two out of the three total results are greater or equal to LLN), at screening. Where there is a clear diurnal effect on the result participants may be included if variations are considered not clinically relevant by the Investigator.
33. Current or recurrent disease (e.g., cardiovascular, haematological, neurological, endocrine, immunological, renal, hepatic or gastrointestinal or other conditions, including cholecystectomy or gastrectomy) that could affect the action, absorption, distribution, metabolism or excretion of PQP or could affect clinical assessments or clinical laboratory evaluations.
34. Current or relevant history of physical or psychiatric illness that are not stable or may require a change in treatment, or use of prohibited therapies during the trial,that make the participant unlikely to fully comply with the requirements of the trial or to complete the trial, or any condition that presents undue risk from the investigational product or trial procedures.
35. Any other abnormal findings on vital signs, ECG, physical examination or laboratory assessments that the Investigator judges as likely to interfere with the trial or pose an additional risk in participating.
36. Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participant at risk because of participation in the trial, or may influence the result of the trial or the participant's ability to participate in the trial.
37. Any conditions which in the opinion of the Investigator would make the participant unsuitable for enrolment or could interfere with the participation in or completion of the trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-08-14 (Actual); Primary Completion 2023-12-06 (Actual); Study Completion 2024-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Florence A Milando, MD, MPH, Principal Investigator — Ifakara Health Institute (IHI), Tanzania; Said A Jongo, MD, MMed, PhD, Study Director — Ifakara Health Institute (IHI), Tanzania
Locations (1):
- Ifakara Health Institute (IHI), Bagamoyo Research and Training Centre (BRTC), Bagamoyo, Bagamoyo District, Pwani Region, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
De-Identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available within 6 months after study completion.
Access Criteria: Requestors will be required to sign a Data Access Agreement.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between July 2023 and December 2023 from the local population residing within and surrounding areas of Bagamoyo town in Tanzania. The first participant was screened on 24 July 2023, the first was dosed on 14 August 2023, and the last was dosed on 06 December 2023.
Pre-assignment Details: Of 143 screened participants, 60 met inclusion criteria and were randomised to treatment. For Part 1 (Fasted) 24: Group 1 = 12 and Group 2 = 12. For Part 2 (Fed) 36: Group 3 = 12; Group 4 = 12 and Group 5 = 12
Groups:
- Part 1 (Fasted) : Group 1 Piperaquine Hard Tablet: Participants received a single oral dose of Piperaquine hard tablet, 320mg, administered in a fasting condition of at least 10 hours. (N=12)
  Piperaquine: Piperaquine tetraphosphate hard tablet 320 mg
- Part 1 (Fasted): Group 2: Piperaquine Dispersible Granules: Participants received a single oral dose of Piperaquine dispersible granules 320mg in a fasting condition of at least 10 hours (N=12)
  Piperaquine: Piperaquine tetraphosphate dispersible granules 320mg
- Part 2 Piperaquine Dispersible Granules (Fed): Group 3: High-fat Meal: Participants received a single oral dose of Piperaquine dispersible granules 320mg in fed conditions with a high-fat meal.
  Piperaquine: Piperaquine tetraphosphate dispersible granules 320mg
- Part 2 Piperaquine Dispersible Granules (Fed): Group 4: Low-fat Meal Representative of African Diet.: Participants received a single oral dose of Piperaquine dispersible granules 320mg in fed conditions with a low-fat meal representative of African diet.
  Piperaquine: Piperaquine tetraphosphate dispersible granules 320mg
- Part 2 Piperaquine Dispersible Granules (Fed): Group 5: Whole Milk 250 mL: Participants received a single oral dose of Piperaquine dispersible granules 320mg in fed conditions with 250mL of whole milk.
  Piperaquine: Piperaquine tetraphosphate dispersible granules 320mg
Period: Part 1: Fasted
Arm/Group | Part 1 (Fasted) : Group 1 Piperaquine Hard Tablet | Part 1 (Fasted): Group 2: Piperaquine Dispersible Granules | Part 2 Piperaquine Dispersible Granules (Fed): Group 3: High-fat Meal | Part 2 Piperaquine Dispersible Granules (Fed): Group 4: Low-fat Meal Representative of African Diet. | Part 2 Piperaquine Dispersible Granules (Fed): Group 5: Whole Milk 250 mL
Started | 12 | 12 | 0 | 0 | 0
Completed | 12 | 12 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Part 2: Fed
Arm/Group | Part 1 (Fasted) : Group 1 Piperaquine Hard Tablet | Part 1 (Fasted): Group 2: Piperaquine Dispersible Granules | Part 2 Piperaquine Dispersible Granules (Fed): Group 3: High-fat Meal | Part 2 Piperaquine Dispersible Granules (Fed): Group 4: Low-fat Meal Representative of African Diet. | Part 2 Piperaquine Dispersible Granules (Fed): Group 5: Whole Milk 250 mL
Started | 0 | 0 | 12 | 12 | 12
Completed | 0 | 0 | 12 | 12 | 12
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Part 1 (Fasted) 24 participants: Group 1 = 12; Group 2 = 12 Part 2 (Fed) 36 Participants: Group 3 = 12; Group 4 = 12; Group 5 = 12
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 (Fasted) : Group 1 Piperaquine Hard Tablet | Part 1 (Fasted): Group 2: Piperaquine Dispersible Granules | Part 2 Piperaquine Dispersible Granules (Fed): Group 3: High-fat Meal | Part 2 Piperaquine Dispersible Granules (Fed): Group 4: Low-fat Meal Representative of African Diet. | Part 2 Piperaquine Dispersible Granules (Fed): Group 5: Whole Milk 250 mL | Total
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 60
Age, Categorical [Count of Participants; unit: Participants] — Population: Part 1 (Fasted) 24 participants: Group 1 = 12; Group 2 = 12 Part 2 (Fed) 36 Participants: Group 3 = 12; Group 4 = 12; Group 5 = 12
  Participants
    Part 1 (Fasted): number analyzed (Participants) | 12 | 12 | 0 | 0 | 0 | 24
    Part 1 (Fasted): <=18 years | 0 | 0 |  |  |  | 0
    Part 1 (Fasted): Between 18 and 65 years | 12 | 12 |  |  |  | 24
    Part 1 (Fasted): >=65 years | 0 | 0 | 0 | 0 | 0 | 0
    Part 2 (Fed): number analyzed (Participants) | 0 | 0 | 12 | 12 | 12 | 36
    Part 2 (Fed): <=18 years |  |  | 0 | 0 | 0 | 0
    Part 2 (Fed): Between 18 and 65 years |  |  | 12 | 12 | 12 | 36
    Part 2 (Fed): >=65 years |  |  | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Part 1 (Fasted) 24 participants: Group 1 = 12; Group 2 = 12 Part 2 (Fed) 36 Participants: Group 3 = 12; Group 4 = 12; Group 5 = 12
  years
    Part 1 (Fasted): number analyzed (Participants) | 12 | 12 | 0 | 0 | 0 | 24
    Part 1 (Fasted) | 29.1 (6.24) | 28.3 (4.74) |  |  |  | 28.7 (5.43)
    Part 2 (Fed): number analyzed (Participants) | 0 | 0 | 12 | 12 | 12 | 36
    Part 2 (Fed) |  |  | 28.2 (7.02) | 28.6 (8.15) | 32.4 (10.14) | 29.7 (8.51)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Part 1 (Fasted) 24 participants: Group 1 = 12; Group 2 = 12 Part 2 (Fed) 36 Participants: Group 3 = 12; Group 4 = 12; Group 5 = 12
  Participants
    Part 1 (Fasted): number analyzed (Participants) | 12 | 12 | 0 | 0 | 0 | 24
    Part 1 (Fasted): Female | 7 | 4 |  |  |  | 11
    Part 1 (Fasted): Male | 5 | 8 |  |  |  | 13
    Part 2 (Fed): number analyzed (Participants) | 0 | 0 | 12 | 12 | 12 | 36
    Part 2 (Fed): Female |  |  | 6 | 7 | 6 | 19
    Part 2 (Fed): Male |  |  | 6 | 5 | 6 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Part 1 (Fasted) 24 participants: Group 1 = 12; Group 2 = 12 Part 2 (Fed) 36 Participants: Group 3 = 12; Group 4 = 12; Group 5 = 12
  Participants
    Part 1 (Fasted): number analyzed (Participants) | 12 | 12 | 0 | 0 | 0 | 24
    Part 1 (Fasted): American Indian or Alaska Native | 0 | 0 |  |  |  | 0
    Part 1 (Fasted): Asian | 0 | 0 |  |  |  | 0
    Part 1 (Fasted): Native Hawaiian or Other Pacific Islander | 0 | 0 |  |  |  | 0
    Part 1 (Fasted): Black or African American | 12 | 12 |  |  |  | 24
    Part 1 (Fasted): White | 0 | 0 |  |  |  | 0
    Part 1 (Fasted): More than one race | 0 | 0 |  |  |  | 0
    Part 1 (Fasted): Unknown or Not Reported | 0 | 0 |  |  |  | 0
    Part 2 (Fed): number analyzed (Participants) | 0 | 0 | 12 | 12 | 12 | 36
    Part 2 (Fed): American Indian or Alaska Native |  |  | 0 | 0 | 0 | 0
    Part 2 (Fed): Asian |  |  | 0 | 0 | 0 | 0
    Part 2 (Fed): Native Hawaiian or Other Pacific Islander |  |  | 0 | 0 | 0 | 0
    Part 2 (Fed): Black or African American |  |  | 12 | 12 | 12 | 36
    Part 2 (Fed): White |  |  | 0 | 0 | 0 | 0
    Part 2 (Fed): More than one race |  |  | 0 | 0 | 0 | 0
    Part 2 (Fed): Unknown or Not Reported |  |  | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Tanzania | 12 | 12 | 12 | 12 | 12 | 60
Body Mass Index (BMI) [Mean (Standard Deviation); unit: units on a scale (kg/m^2)] — Population: Part 1 (Fasted) 24 participants: Group 1 = 12; Group 2 = 12 Part 2 (Fed) 36 Participants: Group 3 = 12; Group 4 = 12; Group 5 = 12
  units on a scale (kg/m^2)
    Part 1 (Fasted): number analyzed (Participants) | 12 | 12 | 0 | 0 | 0 | 24
    Part 1 (Fasted) | 22.127 (3.3784) | 21.355 (3.0850) |  |  |  | 21.741 (3.1884)
    Part 2 (Fed): number analyzed (Participants) | 0 | 0 | 12 | 12 | 12 | 36
    Part 2 (Fed) |  |  | 23.434 (3.7032) | 22.853 (3.3968) | 22.540 (3.6998) | 22.943 (3.5185)

OUTCOME MEASURES:

1. Primary Outcome: Relative Bioavailability (Frel) of the Maximum Observed Plasma Concentration (Cmax) of the PQP Dispersible Granule Compared to the PQP Hard Tablet in the Fasted State (Frel Cmax).
Description: Blood samples are analysed for PQP concentrations at the indicated time points to determine the maximum observed plasma concentration (Cmax) for PQP dispersible granule (test) and PQP hard tablet (reference) in the fasted state. Pharmacokinetic parameters are determined using standard non-compartmental analysis. Frel Cmax is calculated as the (%) ratio of Cmax of the PQP dispersible granule compared to the PQP hard tablet in the fasted state.
Time Frame: Plasma samples taken pre-dose -0.5 hours, then 1, 2, 3, 4, 5, 6, 7, 8, 12, 24, 48, Day 5, Day 8, Day 15, Day 22 and Day 30 post-dose.
Population: The PK analysis set included all participants with sufficient plasma samples taken for at least one of the PK variables to be calculated, who received any study treatment and who experienced no protocol deviations with relevant impact on PK data.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Part 1 Group 1 PQP Hard Tablet: Group 1: Piperaquine hard tablet, 320mg (administered in fasting condition of at least 10 hours) (N=12) Piperaquine Phosphate: PQP hard tablet 320 mg; single dose (320 mg) given orally with 240 ml of water
- Part 1: Group 2 PQP Dispersible Granules: Group 2: Piperaquine dispersible granules 320mg administered in fasting condition of at least 10 hours (N=12) Piperaquine Phosphate: PQP dispersible granules 320 mg dose equivalent dispersed in 25 ml of water; single dose (320 mg) given orally
Arm/Group | Part 1 Group 1 PQP Hard Tablet | Part 1: Group 2 PQP Dispersible Granules
Number analyzed (Participants) | 12 | 12
ng/mL | 37.4 (71.46) | 27.6 (61.64)
Statistical Analysis 1: Comparison: Part 1 Group 1 PQP Hard Tablet vs Part 1: Group 2 PQP Dispersible Granules; Test type: Equivalence — The treatment was considered as bioequivalent if the 90% confidence interval (CI) for geometric least square mean ratios (GMR) of Cmax falls within the acceptance range of 80.00 % to 125.00 %; geometric least square mean ratios (GMR) = 73.9, 90% CI 2-sided [48.32 to 113.02]

2. Primary Outcome: Relative Bioavailability (Frel) of the Area Under the Plasma Concentration-time Curve From Time Zero to 72h Hours (AUC0-72h) of the PQP Dispersible Granule Compared to the PQP Hard Tablet in the Fasted State (Frel AUC0-72h).
Description: Blood samples are analysed for PQP concentrations at the indicated time points to calculate the area under the plasma concentration-time curve from time zero to 72 hours (AUC0-72h) for PQP dispersible granule (test) and PQP hard tablet (reference) in the fasted state. Pharmacokinetic parameters are determined using standard non-compartmental analysis. Frel AUC0-72h is calculated as the ratio of AUC0-72h of the PQP dispersible granule compared to the PQP hard tablet in the fasted state.
Time Frame: as for outcome 1
Population: The PK analysis set included all participants who had sufficient plasma samples taken for at least one of the PK variables to be calculated and who received any study treatment and experienced no protocol deviations with relevant impact on PK data.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Group 1 PQP Hard Tablet: Group 1: Piperaquine hard tablet, 320mg (administered in fasting condition of at least 10 hours) (N=12) Piperaquine Phosphate: PQP hard tablet 320 mg; single dose (320 mg) given orally with 240 ml of water
- Group 2: Piperaquine Dispersible Granules: Group 2: Piperaquine dispersible granules 320mg administered in fasting condition of at least 10 hours (N=12) Piperaquine Phosphate: PQP dispersible granules 320 mg dose equivalent dispersed in 25 ml of water; single dose (320 mg) given orally
Arm/Group | Group 1 PQP Hard Tablet | Group 2: Piperaquine Dispersible Granules
Number analyzed (Participants) | 12 | 12
ng*h/mL | 809.7 (42.77) | 610.6 (43.41)
Statistical Analysis 1: Comparison: Group 1 PQP Hard Tablet vs Group 2: Piperaquine Dispersible Granules; Test type: Equivalence — The treatment was considered as bioequivalent if the 90% confidence interval (CI) for geometric least square mean ratios (GMR) of ln-transformed parameters falls within the acceptance range of 80.00 % to 125.00 %; geometric least square mean ratio (GMR) = 75.41, 90% CI 2-sided [56.46 to 100.71]

3. Primary Outcome: Relative Bioavailability (Frel) of the Area Under the Plasma Concentration-time Curve From Time Zero to the Last Quantifiable Concentration (AUC0-t) of the PQP Dispersible Granule Compared to the PQP Hard Tablet in the Fasted State (Frel AUC0-t).
Description: Blood samples are analysed for PQP concentrations at the indicated time points to calculate the area under the plasma concentration-time curve from time zero to the last quantifiable concentration (AUC0-t) for PQP dispersible granule (test) and PQP hard tablet (reference) in the fasted state. Pharmacokinetic parameters are determined using standard non-compartmental analysis. Frel AUC0-t is calculated as the ratio of AUC0-t of the PQP dispersible granule compared to the PQP hard tablet in the fasted state.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Group 1 PQP Hard Tablet | Group 2: Piperaquine Dispersible Granules
Number analyzed (Participants) | 12 | 12
ng*h/mL | 3267.1 (31.74) | 2824.3 (37.84)
Statistical Analysis 1: Comparison: Group 1 PQP Hard Tablet vs Group 2: Piperaquine Dispersible Granules; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; geometric least square mean ratios (GMR) = 86.45, 90% CI 2-sided [68.16 to 109.63]

4. Primary Outcome: Relative Bioavailability (Frel) of the Area Under the Plasma Concentration-time Curve From Time Zero to 168 Hours (AUC0-168h) of the PQP Dispersible Granule Compared to the PQP Hard Tablet in the Fasted State (Frel AUC0-168h.
Description: Blood samples are analysed for PQP concentrations at the indicated time points to calculate the area under the plasma concentration-time curve from time zero to 168 hours (AUC0-168h) for PQP dispersible granule (test) and PQP hard tablet (reference) in the fasted state. Pharmacokinetic parameters are determined using standard non-compartmental analysis. Frel AUC0-168h is calculated as the ratio of the AUC0-168h of the PQP dispersible granule compared to the PQP hard tablet in the fasted state.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Group 1 PQP Hard Tablet | Group 2: Piperaquine Dispersible Granules
Number analyzed (Participants) | 12 | 12
ng*h/mL | 1373.1 (36.53) | 1066.5 (42.2)
Statistical Analysis 1: Comparison: Group 1 PQP Hard Tablet vs Group 2: Piperaquine Dispersible Granules; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; geometric least square mean ratios (GMR) = 77.67, 90% CI 2-sided [59.49 to 101.39]

5. Primary Outcome: Relative Bioavailability (Frel) of the Area Under the Plasma Concentration-time Curve From Time Zero Extrapolated to Infinity (AUC0-∞) of the PQP Dispersible Granule Compared to the PQP Hard Tablet in the Fasted State (Frel AUC0-∞).
Description: Blood samples are analysed for PQP concentrations at the indicated time points to calculate the area under the plasma concentration-time curve from time zero extrapolated to infinity (AUC0-∞) for PQP dispersible granule (test) and PQP hard tablet (reference) in the fasted state. Pharmacokinetic parameters are determined using standard non-compartmental analysis. Frel AUC0-∞ is calculated as the ratio of the AUC0-∞ of the PQP dispersible granule compared to the PQP hard tablet in the fasted state.
Time Frame: Plasma samples taken pre-dose 0.5 hours, then 1, 2, 3, 4, 5, 6, 7, 8, 12, 24, 48, Day 5, Day 8, Day 15, Day 22 and Day 30 post-dose.
Population: The PK analysis set included all participants who had sufficient plasma samples taken for at least one of the PK variables to be calculated and who received any study treatment and experienced no protocol deviations with relevant impact on PK data. The AUC0-inf was reliably determined (extrapolation to infinity was <20%) for only one participant in the Test group and two participants in the Reference group/
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Group 1 PQP Hard Tablet | Group 2: Piperaquine Dispersible Granules
Number analyzed (Participants) | 2 | 1
ng*h/mL | 4597.8 (29.25) | 2539.7
Statistical Analysis 1: Comparison: Group 1 PQP Hard Tablet vs Group 2: Piperaquine Dispersible Granules; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; geometric least square mean ratios (GMR) = 55.24, 90% CI 2-sided [6.03 to 113.02] — For AUC0-inf, the GMR and 90% CI values were unreliable as there was only 1 calculable value for the Test (Group 2) and 2 values for the Reference (Group 1) products

ADVERSE EVENTS:
Time Frame: The investigator was responsible for documenting and reporting all AEs occurring in the clinical trial. The period of observation for the collection of AEs extended from the time of signing consent to the final visit, a maximum of 75 days. All AEs were recorded until the end of the study. All SAEs which came to the attention of the Investigator within 30 days from the end of the study treatment were also recorded.
Description: * Pre-treatment adverse event: AEs between informed consent and Investigational Medicinal Product administration.
  * Adverse Event: Any unfavourable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of a medicinal product, whether or not considered related to it.
  * TEAEs: An event that emerges during treatment, have been absent pre-treatment or worsens relative to the pre-treatment state.
Groups:
- Part 1 (Fasted): Group 1: Piperaquine Hard Tablets: Participants received a single oral dose of Piperaquine hard tablets 320mg (administered in fasting condition of at least 10 hours) (N=12)
  Piperaquine: Piperaquine tetraphosphate hard tablets 320mg
  Piperaquine Tetraphosphate uncoated tablets: Piperaquine tetraphosphate hard tablet 320 mg; single dose (320 mg) given orally with 240 ml of water
- Part 1 (Fasted): Group 2: Piperaquine Dispersible Granules: Participants received a single oral dose of Piperaquine dispersible granule 320mg (administered in fasting condition of at least 10 hours) (N=12)
  Piperaquine: Piperaquine tetraphosphate dispersible granules 320mg
  Piperaquine Tetraphosphate dispersible granules: Piperaquine tetraphosphate dispersible granules 320 mg dose equivalent dispersed in 25 ml of water; single dose (320 mg) given orally
- Part 2 (Fed): Group 3: Piperaquine Dispersible Granules: Participants received a single oral dose of Piperaquine dispersible granule 320mg administered with a high-fat meal (N=12)
  Piperaquine: Piperaquine tetraphosphate dispersible granules 320mg
  Piperaquine Tetraphosphate dispersible granules: Piperaquine tetraphosphate dispersible granules 320 mg dose equivalent dispersed in 25 ml of water; single dose (320 mg) given orally
- Part 2 (Fed): Group 4: Piperaquine Dispersible Granules: Participants received a single oral dose of Piperaquine dispersible granule 320mg administered with a low-fat meal representative of African diet. (N=12)
  Piperaquine: Piperaquine tetraphosphate dispersible granules 320mg
  Piperaquine Tetraphosphate dispersible granules: Piperaquine tetraphosphate dispersible granules 320 mg dose equivalent dispersed in 25 ml of water; single dose (320 mg) given orally
- Part 2 (Fed): Group 5: Piperaquine Dispersible Granules: Participants received a single oral dose of Piperaquine dispersible granule 320mg administered with whole milk (250ml) (N=12)
  Piperaquine: Piperaquine tetraphosphate dispersible granules 320mg
  Piperaquine Tetraphosphate dispersible granules: Piperaquine tetraphosphate dispersible granules 320 mg dose equivalent dispersed in 25 ml of water; single dose (320 mg) given orally
Arm/Group | Part 1 (Fasted): Group 1: Piperaquine Hard Tablets | Part 1 (Fasted): Group 2: Piperaquine Dispersible Granules | Part 2 (Fed): Group 3: Piperaquine Dispersible Granules | Part 2 (Fed): Group 4: Piperaquine Dispersible Granules | Part 2 (Fed): Group 5: Piperaquine Dispersible Granules
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 1/12 | 1/12 | 0/12 | 1/12 | 0/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 (Fasted): Group 1: Piperaquine Hard Tablets (N=12) | Part 1 (Fasted): Group 2: Piperaquine Dispersible Granules (N=12) | Part 2 (Fed): Group 3: Piperaquine Dispersible Granules (N=12) | Part 2 (Fed): Group 4: Piperaquine Dispersible Granules (N=12) | Part 2 (Fed): Group 5: Piperaquine Dispersible Granules (N=12)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Participant# 122, results for all collected samples were below the lower limit of quantification (LLOQ) and no PK parameters could be generated. So, data from Participant# 122 was not included in the summary statistics.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol (2023-11-08): https://cdn.clinicaltrials.gov/large-docs/82/NCT05930782/Prot_000.pdf
  • Statistical Analysis Plan: Pharmacokinetic Data Analysis Plan (2023-10-02): https://cdn.clinicaltrials.gov/large-docs/82/NCT05930782/SAP_001.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan (2023-12-19): https://cdn.clinicaltrials.gov/large-docs/82/NCT05930782/SAP_002.pdf
  • Informed Consent Form (2023-02-14): https://cdn.clinicaltrials.gov/large-docs/82/NCT05930782/ICF_003.pdf